CLINICAL TRIAL: NCT05953896
Title: Efficacy of Hyaluronic Acid Gel Injection Versus Multilayer Leukocyte Platelet Rich Fibrin (L-PRF) in The Interdental Papilla Reconstruction: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of HA Gel Injection Versus Multilayer (L-PRF) in the Interdental Papilla Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Elleithy (Other)
Responsible Party: Sponsor-Investigator, Aya Elleithy, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDASU-REC 012112
Record Dates: First submitted 2023-03-17; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Gingival Papillary Cratering
Keywords: interdental papilla; multilayer L-PRF; Hyaluronic acid gel

STUDY DESIGN:
Intervention Model Description: this study is designed as a parallel randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid gel (Experimental): will include 10 patients undergoing non invasive reconstruction of interdental papilla using injectable Hyaluronic acid gel
  Interventions: Combination Product: Hyaluronic acid gel
- Multilayer L-PRF (Active Comparator): will include 10 patients undergoing minimally invasive surgery for reconstruction of interdental papilla using multilayer L-PRF membranes
  Interventions: Combination Product: Multilayer L-PRF membranes

INTERVENTIONS:
Combination Product: Hyaluronic acid gel — For the Hyaluronic acid gel group: HA gel was injected 2-3mm apical to the coronal tip of the involved papillae and the needle was directed coronally with an angulation of 45° to the long axis of the tooth, and the bevel directed apically until papilla became blanched. The injection was given at each papilla at the following intervals baseline, one week and two weeks.
  Other Names: HA gel
  Arms: Hyaluronic acid gel
Combination Product: Multilayer L-PRF membranes — For the multilayer L-PRF group: A single semilunar incision is made in the buccal vestibule, apical to the muco-gingival junction in the mid interproximal area of the papilla to be treated.Tunneling of the incisions has maintained the full height and thickness of the gingiva. Multilayer L-PRF membranes were prepared according to Pinto's protocol immediately prior to the surgery and placed in the tunnel then incision was closed with simple interrupted sutures.
  Arms: Multilayer L-PRF

SUMMARY:
This research aims to investigate the effectiveness of non invasive application Hyaluronic acid gel injection versus minimally invasive surgical approach using multilayer L-PRF both clinically and radiographically as a suitable treatment modality for interdental papillary deficiency.

DETAILED DESCRIPTION:
A total of 20 patients recruited from the outpatient clinic of Oral Medicine, Periodontology and Oral Diagnosis department, Faculty of Dentistry, Ain-Shams University and seeking treatment for black triangles for esthetic reason. Patients meeting the eligibility criteria are equally and randomly allocated in two different groups. group one Included 10 patients who received interdental papillary reconstruction using multiple layers of L-PRF. Group two Included 10 patients who received interdental papillary reconstruction using Hyaluronic acid gel injection. In the follow-up phase, patients were recalled after 3 and 6 months from intervention where clinical re-measurement of the black triangles and standardized digital clinical photographs and radiographs are done. Black triangle height and surface area was measured and other clinical parameters (Modified papillary bleeding index, Gingival index, clinical attachment level and periodontal probing depth) were assessed at baseline, 3 months and 6 months periods. patient satisfaction was evaluated using the patient satisfaction questionnaire (PSQ-18, short form) at baseline. pain and discomfort was evaluated using Numerical rating scale (NRS) at baseline, 3 months and 6 months periods. Global esthetic improvement scale (GAIS) was evaluated at 3 months and 6 months periods.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders aged from 18-45 years.
2. Systemically healthy patients.
3. Patients with IDP loss class I or II of esthetic zone in upper and lower anterior and premolar teeth according to Nordland and Tarnow's classification (Class I: Presence of the tip of the papilla between interdental contact point and the interproximal CEJ)
4. Presence of sufficient interdental alveolar bone (i.e. the vertical distance from the interdental contact point to the crest of the interdental bone is ≥ 5 mm) that was confirmed clinically by bone sounding.
5. A band of keratinized tissue should be present around the test teeth ≥ 2 mm
6. Periodontal phenotype of the area to be treated is ≥ 2 mm in thickness. Surgical reconstruction of IDP is influenced by gingival tissue phenotype, outcome of papilla reconstruction is better in cases with a thick gingival unit
7. Patients with good oral hygiene and caring about esthetics and concerned to go through the management of "black triangles" by interdental papillae reconstruction in esthetic zone.

Exclusion criteria:

1. Teeth with acute periapical pathosis.
2. Patients with poor oral hygiene, incompliance to treatment and persistence of gingival inflammation after phase I therapy.
3. Pregnant and lactating females.
4. Patients having para-functional habits or local causes as, malocclusion, interdental spacing, rotation, inclination or crowding.
5. Smokers, alcoholics or drug abusers.
6. Vulnerable group of patients, orphans, handicapped, prisoners or mentally retarded patients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The gingival black triangle height | six months
  to evaluate the influence of hyaluronic acid gel injection versus multilayer L-PRF on the height of black triangle

SECONDARY OUTCOMES:
Assessment pf patient satisfaction using Patient Satisfaction Questionnaire | patients scores are evaluated at baseline immediately after the procedure
  evaluation of patient satisfaction using patient Satisfaction questionnaire (PSQ-18, short form), patients are informed to fill and sign the questionnaire with 18 questions to evaluate their satisfaction of the recieved intervention
Post operative pain assessment using Numerical Pain Rating Scale | six months
  To evaluate patient's perception of postoperative pain during the treatment time using the NRS (Numeric Pain Rating Scale). The NRS is an 11-point numeric scale that ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Assessment of esthetic appearance using the GAIS (global esthetic improvement scale) | six months
  patients satisfaction of their esthetic appearance will be rocorded using the global esthetic improvement scale with ranges (1: worsened) (2: unchanged) (3: improved) (4: much improved)

CONTACTS AND LOCATIONS:
Overall Officials: Aya Alleithy, teaching assistant, Principal Investigator — Teaching assistant at Department of Oral medicine, Periodontology, and Oral Diagnosis, Faculty of Dentistry, A; Hala Abu El-Ela, proffessor, Study Director — Professor of Oral Medicine, Periodontology and Oral Diagnosis , Faculty of Dentistry-Ain Shams University & Misr International university; Susan Sarhan, lecturer, Study Director — Lecturer of Oral Medicine and Periodontology and Oral diagnosis, Faculty of Dentistry, Ain Shams University
Locations (1):
- faculty of Dentistry. Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No